CLINICAL TRIAL: NCT03558607
Title: Concomitant Ruxolitinib Induction and Maintenance With Cytarabine Based Chemotherapy in Secondary Acute Myelogenous Leukemia Evolving From Myeloproliferative Neoplasm
Brief Title: The Role of Ruxolitinib in Secondary Acute Myelogenous Leukemia Evolving From Myeloproliferative Neoplasm
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1803-145-934
Record Dates: First submitted 2018-05-24; First posted 2018-06-15 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Secondary Acute Myelogenous Leukemia Evolving From Myeloproliferative Disorder
MeSH Terms: interventions — ruxolitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental)
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Induction chemotherapy include combination of cytarabine (200mg/m2) and idarubicin (12mg/m2). Both 7+3 and 5+2 regimen is allowed according to age and performance status (PS) as follows;
  * If Age < 55 years and ECOG PS < 2 : 7+3 regimen
  * If Age ≥ 55 years or ECOG PS = 2 : 5+2 regimen
  Ruxolitinib is administered for 14 days during induction/consolidation phase. After complete remission after induction, ruxolitinib is administered for the first 14 days during consolidation chemotherapy. Maximum 3 cycles of consolidation is recommended. In case of allogeneic stem cell transplantation (alloSCT), ruxolitinib is discontinued at the time of transplantation. After completion of consolidation, 2 years of ruxolitinib maintenance is planned. The follow-up period is from the time of enrollment until 24 months.

SUMMARY:
This trial aimed to investigate the therapeutic efficacy of ruxolitinib in combination with cytotoxic chemotherapy for post-myeloproliferative neoplasm secondary acute myeloid leukemia.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is an uncommon, but often deadly complication of myeloproliferative neoplasms (MPN). Post-MPN AML is aggressive and resistant to conventional treatment with median survival of 3-5 months. Although allogeneic stem cell transplantation (alloSCT) have some prospective of promise in these patient, most of them are ineligible for alloSCT because of advanced age at diagnosis, comorbidities and scarcity of a compatible donor. Therefore, there is an urgent need for new therapeutic strategy for post-MPN AML.

Cytogenetic and/or molecular abnormalities associated with poor prognosis are quite common in patients with post-MPN AML. Although these findings likely contribute to the aggressive natural history and resistance to standard therapies, the genetic complexity of post-MPN AML may ultimately permit targeted therapy. Among these abnormalities, Janus kinase 2 (JAK2) has come to the fore recently. JAK2 V617F mutation, which is a hallmark of MPN, has been reported to be carried in approximately 35-50% of patients with post-MPN AML. We believe that this mutation be the most oncogenic driver in post-MPN AML.

In fact, BCR/ABL(+) acute leukemia (either blast crisis of CML or Ph+ ALL) is a similar disease model of the post-MPN AML. The clinical outcome of these disease has improved dramatically with ABL tyrosine kinase inhibitors (TKIs), such as imatinib, and nilotinib. It is a standard practice to give ABL TKI along with cytotoxic chemotherapy to BCR/ABL(+) acute leukemia. On the other hand, in BCR/ABL(+) acute leukemia, it is well known that single agent ABL TKI is not sufficient to control disease.

Likewise, ruxolitinib, which is a targeted agent for JAK2, have a great possibility to show efficacy for post-MPN AML when combined with cytotoxic agents. In a previous investigational study of ruxolitinib for refractory/relapsed leukemias, 2 of 3 AML patients evolving from MPN achieved complete remission with two cycles of ruxolitinib. In fact, many clinical trials are ongoing to investigate the therapeutic efficacy of ruxolitinib in post-MPN AML as a single agent.

However, considering a lesson from BCR/ABL(+) acute leukemia, ruxolitinib as a single agent may not be enough to cure these patients with post-MPN AML. Hence, for patients who are fit for intensive chemotherapy, it would easily conjectured that ruxolitinib in combination with cytotoxic chemotherapy would be better for these patients. Therefore, combination of ruxolitinib and cytotoxic chemotherapy would be an optimal treatment for post-MPN AML. From an epidemiologic perspective, it is true that post-MPN AML develops in elderly patients frequently. However, patients who fit for intensive chemotherapy are also encountered in the clinic for post-MPN AML not infrequently, justifying this study design. NCCN guideline also recommend intensive induction treatment for patients > 60 years when there performance and comorbidity allows intensive treatment.

In this study, the therapeutic efficacy of ruxolitinib in combination with cytotoxic chemotherapy for post-MPN AML will be investigated. Unlike other clinical trials induction and consolidation treatment should include cytotoxic chemotherapeutic agents in addition to ruxolitinib.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically confirmed AML following MPN
* ECOG performance status 2 or better
* Adequate physical condition that could tolerate cytotoxic induction chemotherapy judged by investigator
* Age 18 years or older
* Adequate cardiac function
* Adequate hepatic, and renal function
* Serum creatinine ≤ 2.5 mg/dl
* ALT (SGOT) and/or AST (SGPT) equal to or than 1.5 x upper limit of normal
* Life expectancy of ≥ 3 months
* Signed and dated informed consent of document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment
* For women of childbearing age, it should be confirmed that they are not pregnant and that they should be contraception during the study period and for up to 4 weeks after the end of the study
* Male should agree to the barrier method during the study period and up to four weeks after the end of the study

Exclusion Criteria:

* Diagnosis of any serious secondary malignancy within the last 2 years, except for adequately treated basal cell or squamous cell carcinoma of skin, or in situ carcinoma of cervix uteri
* Pregnancy or breast feeding
* Other severe acute or chronic medical or psychiatric condition
* Prior treatment with ruxolitinib
* Patients who received other chemotherapy within 2 weeks of the study enrollment
* Patients participating in other clinical studies at the time of registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2018-05-17 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
complete remission rate | After 12 months from induction chemotherapy
complete remission with incompletre recovery rate | After 12 months from induction chemotherapy

SECONDARY OUTCOMES:
Overall survival | 3, 6, 12, 24 months after induction chemotherapy
  from the date of transplantation to death from any cause
Progression-free survival | 3, 6, 12, 24 months after induction chemotherapy
  from the date of transplantation to the date of disease progression or death from any cause
Toxicity profile | 3, 6, 12, 24 months after induction chemotherapy
  according to CTCAE version 4.03

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdulkarim K, Girodon F, Johansson P, Maynadie M, Kutti J, Carli PM, Bovet E, Andreasson B. AML transformation in 56 patients with Ph- MPD in two well defined populations. Eur J Haematol. 2009 Feb;82(2):106-11. doi: 10.1111/j.1600-0609.2008.01163.x. PMID 19134023
- [Background] Koh Y, Kim I, Bae JY, Song EY, Kim HK, Yoon SS, Lee DS, Park SS, Park MH, Park S, Kim BK. Prognosis of secondary acute myeloid leukemia is affected by the type of the preceding hematologic disorders and the presence of trisomy 8. Jpn J Clin Oncol. 2010 Nov;40(11):1037-45. doi: 10.1093/jjco/hyq097. Epub 2010 Jun 29. PMID 20587614
- [Background] Mesa RA, Li CY, Ketterling RP, Schroeder GS, Knudson RA, Tefferi A. Leukemic transformation in myelofibrosis with myeloid metaplasia: a single-institution experience with 91 cases. Blood. 2005 Feb 1;105(3):973-7. doi: 10.1182/blood-2004-07-2864. Epub 2004 Sep 23. PMID 15388582
- [Background] Passamonti F, Rumi E, Arcaini L, Castagnola C, Lunghi M, Bernasconi P, Giovanni Della Porta M, Columbo N, Pascutto C, Cazzola M, Lazzarino M. Leukemic transformation of polycythemia vera: a single center study of 23 patients. Cancer. 2005 Sep 1;104(5):1032-6. doi: 10.1002/cncr.21297. PMID 16047334
- [Background] Tam CS, Nussenzveig RM, Popat U, Bueso-Ramos CE, Thomas DA, Cortes JA, Champlin RE, Ciurea SE, Manshouri T, Pierce SM, Kantarjian HM, Verstovsek S. The natural history and treatment outcome of blast phase BCR-ABL- myeloproliferative neoplasms. Blood. 2008 Sep 1;112(5):1628-37. doi: 10.1182/blood-2008-02-138230. Epub 2008 Jun 19. PMID 18566326
- [Background] Cherington C, Slack JL, Leis J, Adams RH, Reeder CB, Mikhael JR, Camoriano J, Noel P, Fauble V, Betcher J, Higgins MS, Gillette-Kent G, Tremblay LD, Peterson ME, Olsen JJ, Tibes R, Mesa RA. Allogeneic stem cell transplantation for myeloproliferative neoplasm in blast phase. Leuk Res. 2012 Sep;36(9):1147-51. doi: 10.1016/j.leukres.2012.04.021. Epub 2012 May 11. PMID 22578777
- [Background] Heaney ML, Soriano G. Acute myeloid leukemia following a myeloproliferative neoplasm: clinical characteristics, genetic features and effects of therapy. Curr Hematol Malig Rep. 2013 Jun;8(2):116-22. doi: 10.1007/s11899-013-0154-5. PMID 23572311
- [Background] Abdel-Wahab O, Manshouri T, Patel J, Harris K, Yao J, Hedvat C, Heguy A, Bueso-Ramos C, Kantarjian H, Levine RL, Verstovsek S. Genetic analysis of transforming events that convert chronic myeloproliferative neoplasms to leukemias. Cancer Res. 2010 Jan 15;70(2):447-52. doi: 10.1158/0008-5472.CAN-09-3783. Epub 2010 Jan 12. PMID 20068184
- [Background] Beer PA, Delhommeau F, LeCouedic JP, Dawson MA, Chen E, Bareford D, Kusec R, McMullin MF, Harrison CN, Vannucchi AM, Vainchenker W, Green AR. Two routes to leukemic transformation after a JAK2 mutation-positive myeloproliferative neoplasm. Blood. 2010 Apr 8;115(14):2891-900. doi: 10.1182/blood-2009-08-236596. Epub 2009 Dec 11. PMID 20008300
- [Background] Eghtedar A, Verstovsek S, Estrov Z, Burger J, Cortes J, Bivins C, Faderl S, Ferrajoli A, Borthakur G, George S, Scherle PA, Newton RC, Kantarjian HM, Ravandi F. Phase 2 study of the JAK kinase inhibitor ruxolitinib in patients with refractory leukemias, including postmyeloproliferative neoplasm acute myeloid leukemia. Blood. 2012 May 17;119(20):4614-8. doi: 10.1182/blood-2011-12-400051. Epub 2012 Mar 15. PMID 22422826
- [Background] Simon R. Optimal two-stage designs for phase II clinical trials. Control Clin Trials. 1989 Mar;10(1):1-10. doi: 10.1016/0197-2456(89)90015-9. PMID 2702835